CLINICAL TRIAL: NCT00254527
Title: Colonization, Infection, and Molecular Typing of Methicillin-Resistant Staphylococcus Aureus (MRSA) in Children.
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: IRB# 04 11-135E
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2007-05-02 (Estimated); Status verified 2005-11

CONDITIONS: Methicillin Resistance; Staphylococcus Aureus
Keywords: Methicillin Resistant Staphylococcus aureus; Children; Colonization; Risk Factor
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The intent of this study is to:

1. Define the prevalence of MRSA carriage in the pediatric population in Kansas City.
2. Systematically define patient risk factors for MRSA carriage and infection.
3. Characterize the unique genetic characteristics of MRSA strains, both community acquired (CA) and healthcare associated (HCA) that are present in the different pediatric populations.

DETAILED DESCRIPTION:
Staphylococcus aureus (SA) are responsible for both localized and invasive infections including carbuncles, cellulitis, lymph node abscess, and wound infections among others. SA is a ubiquitous environmental organism that colonizes 30-50% adults and more than 50% of children with underlying skin disorders. Hematogenous seeding can result in fulminant infection, and sites as diverse as bone, joint, lung, muscle, pericardium, endocardium, and other vascular structures can be involved. Factors which are known to increase the risk for colonization include the presence of underlying skin disorders and history of frequent needle use which occur in the setting of diabetes, or hemodialysis. Health care workers have traditionally been noted to have higher carriage rates.

MRSA strains emerged in the last two decades in the US and similarities to the evolution of penicillin resistant S. aureus were noted with colonization and infection in the hospital based setting noted first. Again, risk factors for MRSA colonization or infection in the hospital were noted to include prior antibiotic exposure, admission to an intensive care unit, surgery, and exposure to an MRSA-colonized patient. Emergence of CA-MRSA strains has been noted in the last decade having resistance to methicillin and erythromycin but susceptibility to clindamycin. These strains have challenged the practitioner's approach to the treatment of common skin and soft tissue infections as well as the management of invasive disease. The importance of such strains was underscored by the 1999 report detailing the deaths of 4 US children with invasive MRSA infection, none of whom had identifiable MRSA risk factors. Pulsed field typing of the isolates confirmed that these community strains were distinct from nosocomial strains isolated from patients in local hospitals.

This study seeks to more clearly define the prevalence of MRSA carriage; better identify risk factors through personal interview; and further identify resistance patterns and molecular strains. This data will guide physicians at Children's Mercy and in the community at large in choosing the best treatment option for children with MRSA infections.

The absence of traditional risk factors for MRSA infection has been noted in children with CA infections. Many studies that describe risk factors in MRSA patients do so by retrospective review of the medical record. Misclassification of patients may occur as physicians do not routinely document the presence or absence of such risk factors, particularly among household contacts.

This study will look at nasal colonization for 500 children in the Kansas City area to determine prevalence of MRSA colonization. During the study period, all invasive MRSA isolates will also be collected. Pulsed field typing will be done to determine whether the strains are community or healthcare associated and both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

Colonization:

- Children ages 3 months to 12 years

Invasive:

- Invasive MRSA infection

Exclusion Criteria:

Colonization:

-None

Invasive:

-Those without invasive MRSA infection

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 477 (Actual)
Dates: Start 2005-01; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Thorell, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Wadlvogel FA. Staphylococcus aureus. In: Mandell GL, Bennett JE, Dolin R, editors. Principles and Practice of Infectious Diseases. 5th ed. Philadelphia: Churchill Livingstone, 2000. p.2072-3
- [Background] Kirby WM. EXTRACTION OF A HIGHLY POTENT PENICILLIN INACTIVATOR FROM PENICILLIN RESISTANT STAPHYLOCOCCI. Science. 1944 Jun 2;99(2579):452-3. doi: 10.1126/science.99.2579.452. PMID 17798398
- [Background] ROZWADOWSKA-DOWZENKO M, LAMERS H. [Infection by penicillin resistant staphylococci]. Pol Tyg Lek (Wars). 1951 May 7;6(18-19):613-7. No abstract available. Undetermined Language. PMID 14875525
- [Background] Ross S, Rodriguez W, Controni G, Khan W. Staphylococcal susceptibility to penicillin G. The changing pattern among community strains. JAMA. 1974 Aug 19;229(8):1075-7. No abstract available. PMID 4276728
- [Background] Gross-Schulman S, Dassey D, Mascola L, Anaya C. Community-acquired methicillin-resistant Staphylococcus aureus. JAMA. 1998 Aug 5;280(5):421-2. No abstract available. PMID 9701074
- [Background] L'Heriteau F, Lucet JC, Scanvic A, Bouvet E. Community-acquired methicillin-resistant Staphylococcus aureus and familial transmission. JAMA. 1999 Sep 15;282(11):1038-9. doi: 10.1001/jama.282.11.1038. No abstract available. PMID 10493201
- [Background] Centers for Disease Control and Prevention (CDC). Four pediatric deaths from community-acquired methicillin-resistant Staphylococcus aureus - Minnesota and North Dakota, 1997-1999. MMWR Morb Mortal Wkly Rep. 1999 Aug 20;48(32):707-10. PMID 21033181
- [Background] Bartlett PC, Martin RJ, Cahill BR. Furunculosis in a high school football team. Am J Sports Med. 1982 Nov-Dec;10(6):371-4. doi: 10.1177/036354658201000611. PMID 7180958
- [Background] Lindenmayer JM, Schoenfeld S, O'Grady R, Carney JK. Methicillin-resistant Staphylococcus aureus in a high school wrestling team and the surrounding community. Arch Intern Med. 1998 Apr 27;158(8):895-9. doi: 10.1001/archinte.158.8.895. PMID 9570176
- [Background] Thorell E, Jackson MA, Bratcher D, Swanson DS, Selvarangan R. Antimicrobial Resistance of Staphylococcus aureus from Kansas City Children: What is the Appropriate Current Therapy for Pediatric Staphylococcal Infections? 42nd Annual Meeting of Infectious Diseases Society of America, Boston, Sept 30- Oct 3, 2004
- [Background] Chambers HF. The changing epidemiology of Staphylococcus aureus? Emerg Infect Dis. 2001 Mar-Apr;7(2):178-82. doi: 10.3201/eid0702.010204. PMID 11294701
- [Background] Hussain FM, Boyle-Vavra S, Daum RS. Community-acquired methicillin-resistant Staphylococcus aureus colonization in healthy children attending an outpatient pediatric clinic. Pediatr Infect Dis J. 2001 Aug;20(8):763-7. doi: 10.1097/00006454-200108000-00009. PMID 11734738
- [Background] McDougal LK, Steward CD, Killgore GE, Chaitram JM, McAllister SK, Tenover FC. Pulsed-field gel electrophoresis typing of oxacillin-resistant Staphylococcus aureus isolates from the United States: establishing a national database. J Clin Microbiol. 2003 Nov;41(11):5113-20. doi: 10.1128/JCM.41.11.5113-5120.2003. PMID 14605147